CLINICAL TRIAL: NCT04898374
Title: Induction Versus Adjuvant Gemcitabine/Cisplatin in Locally Advanced Non-metastatic Nasopharyngeal Carcinoma: A Randomized Phase III Trial
Brief Title: Induction Versus Adjuvant Gemcitabine/Cisplatin in Locally Advanced Non-metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kuwait Cancer Control Center (Other)
Responsible Party: Principal Investigator, Shereen Issa, Dr Shereen Issa, MD, Kuwait Cancer Control Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNIC-NP
Record Dates: First submitted 2021-05-13; First posted 2021-05-24 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Induction chemotherapy; neoadjuvant; adjuvant; non-metastatic; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Randomised controlled non-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Induction Arm (Experimental): patients will receive three cycles of IC Gemcitabin/Cisplatin followed by radical CRT
  Interventions: Drug: Gemcitabin/cisplatin
- Adjuvant Arm (Active Comparator): Patients will receive radical CRT followed by three cycles of AC Gemcitabin/Cisplatin
  Interventions: Drug: Gemcitabin/cisplatin

INTERVENTIONS:
Drug: Gemcitabin/cisplatin — chemotherapy combination

SUMMARY:
The standard of care for locally advanced nasopharyngeal carcinoma is radical chemoradiation(CRT).Recent advances in radiation techniques and supportive measures resulted in improvemnent of locoregional control and quality of life.However distant failure is still the main challenging reason of poor survival

Addition of systemic therapy to concurrent CRT is widely used and accepted as an option to reduce these failures ,however selection of chemotherapy regimen and timing in relation to CRT is controversial.

Doublet and triplet chemotherapy regimens using cisplatin and 5FU are throughly investigated in this setting.Inspite of significant improvement in disease free survival and overall survival they were poorly tolerated.Hence,minority of patients in the daily practice could tolerate those studied regimens as propsed.

Recently, in multicenter randomized trial, Zhang and his group investigated gemcitabine and cisplatin as induction chemotherapy (ICT) added to CRT.It showed improvement in recurrence free survival and overall survival.More importantly 96.7% of the experimental arm completed the treatment protocol.

This was further confirmed by an updated network of meta analysis by Bongiovanni et al.Again the question of "when" is still valid.Our proposal is to compare tolerable regimen in induction versus adjuvant settings.

DETAILED DESCRIPTION:
Background

Nasopharyngeal carcinoma (NPC) is one of the cancers which shows significant geographic prevalence variation. Worldwide, there were 130,000 new cases in 2018.As a non-endemic region, only 35 new cases were diagnosed in Kuwait in the same year. Nevertheless, it accounts for 1.3% of cancer related mortality in Kuwait.

Radical radiotherapy (RT) is the mainstay treatment of NPC for decades. A high cure rate can be achieved for patients with early-stage. The breakthrough in the management of NPC came with the intergroup study 009 which showed significant improved progression free survival with adding chemotherapy (CTH) to the radiation.

As compared to RT alone, concurrent chemoradiation (CRT), showed significant improvement in 10-year overall survival and progression free survival in meta-analysis of nasopharyngeal carcinoma (MAC-NPC) collaborative group. Addition of systemic therapy to concurrent CRT was the proposed solution to treatment failures; whether in the induction (ICT) or adjuvant (ACT) settings. However, ICT or ACT in NPC remains controversial; largely due to inconsistent results of several prospective randomized trials.

The above-mentioned MAC-NPC group reviewed six clinical trials in which CRT followed by ACT was compared with RT alone (administrated without concurrent or adjuvant chemotherapy). Overall survival (OS) was significantly improved compared with RT alone (10-year overall survival 57% versus 43.1%, HR 0.65, 95% CI 0.56-0.76), as well as 10-year progression-free survival; PFS (53.2% versus 38.5%).

However, this was not consistent in endemic areas with high prevalence of Epstein-Barr virus (EBV); which is known causative for NPC. Chen et al reported in a Chinese phase III trial 508 patients with advanced NPC randomized to ACT (cisplatin plus fluorouracil) vs observation following CRT with weekly cisplatin. There was no improvement in the five-year failure-free rate with ACT compared with CRT alone (five-year rate 75% versus 71%, HR 0.88, 95% CI 0.64-1.22) Later, from the same endemic region, Sun Yat-sen university conducted a multi center phase III clinical trial in which 480 patients, stage III to IVB, node-positive NPC were randomly assigned to ICT followed by CRT versus CRT alone. This study showed improvement of recurrence-free survival (RFS) and distant RFS.

Another reason for reluctancy to adopt ICT or ACT in the management of advanced NPC, is the morbidity of current chemotherapy regimens. The high toxicity profile with some of these regimens was the real obstacle toward the use of them. In previous studies, the back bone for adjuvant or induction chemotherapy in NPC has been platinum and 5-fluoruracil, with or without a taxane. This regimen was poorly tolerated, with only 40-60 % of patients could complete their preplanned course of treatment in many trials.

Recently, in multicenter randomized trial, Zhang and his group compared gemcitabine and cisplatin as ICT plus CRT with CRT alone. The 3-year RFS was 85.3% in the induction group and 76.5% in the standard-therapy group (HR 0.51; 95% CI, 0.34 to 0.77; P=0.001). Overall survival at 3 years was 94.6% and 90.3%, respectively (HR 0.43; 95% CI, 0.24 to 0.77). What is more important is that 96.7% of the experimental arm completed 3 cycles of ICT.

On behalf of the Nasopharyngeal Cancer Portal Group of Investigators, Bossi colleagues from Europe, Kuwait, Jordan, Turkey and USA, assessed the impact of treatment intensity within a large retrospective multicenter cohort, nasopharyngeal cancer in non-endemic areas. Our group shared in this pooled analysis and the data showed a higher rate of death and recurrence with non-intensive treatment, (defined as no "added" systemic treatment to CRT).

Ongoing Phase 3 Trials exploring ICT or ACT in NPC:

There are multiple phase 3 trials ongoing to refine the ICT or ACT approach. Sun Yat-sen University is conducting a study comparing TPF with PF as ICT regimen in stage IVa-b NPC (NCT02940925). They also explore the effect of triple combination of ICT, CRT and ACT in high risk NPC (NCT02621970). Another comparison between induction TPF vs adjuvant PF is recruiting (NCT03306121). Fudan University also from China exploring maintenance gemcitabine after radical treatment in N3 disease (NCT03403829). Jiangxi Provincial Cancer Hospital testing adding neoadjuvant and adjuvant PD-1 inhibitor to ICT-CRT (NCT04557020) Another promising strategy to control the distant failures in locally advanced NPC, is to employ immunotherapy in the primary treatment. There are many ongoing trials exploring this strategy, mainly in China. However, the validity in endemic vs non-endemic regions should be taken with caution.

Aim of the study In our proposal we are trying to compare the efficacy and tolerability of ICT followed by CRT with CRT followed ACT in locally advanced NPC

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed Nasopharyngeal carcinoma (according to World Health Organization (WHO) 2. The patient has stage III except T3N0 or IVA disease (according to 8th American Joint Committee on Cancer staging system) 3. WHO performance status 0-1 . 4. The patient must have achieved lawful age to provide informed consent according to local or national law .

  5. Laboratory values performed within 14 days prior to concurrent chemotherapy should be as follows: i) Absolute neutrophil count (ANC) ≥ 1500/mm ii) Platelet count ≥ 100.000/mm iii) Hemoglobin ≥ 8g/dl iv) Urea and serum creatinine ≤ 1.5 mg/dl. (for cisplatin) v) Creatinine clearance ≥ 60 ml/min. (for cisplatin) vi) SGOT and SGPT ≤ 2 × upper limit of laboratory normal 6. Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study therapy

Exclusion Criteria:

1. Age ≥70 or <18
2. The patient has evidence of distant metastatic disease.
3. The patient has received prior systemic chemotherapy within the last three years.
4. The patient has undergone previous surgery for the tumor, other than biopsy.
5. The patient has received prior radiation therapy to the head or neck
6. The patient is pregnant or breast feeding.
7. The patient has a medical (e.g. renal impairment) or psychological condition that would not permit the patient to complete the trial or sign informed consent.
8. Has known history of Human Immunodeficiency Virus (HIV)
9. Has history of a diagnosed and/or treated hematologic or primary solid tumor malignancy,
10. Has a history of severe hypersensitivity reaction to Cisplatin, Gemcitabine or radiotherapy or their analogs
11. Unstable cardiac disease requiring treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Acute and late toxicity assessment | 3-5 years
  Incidence of acute toxicity is calculated for each adverse event respectively, and severity evaluated on based of common terminology criteria for adverse event (CTCAE)
Late radiation toxicity | 5-7 years
  assessed using the radiation therapy oncology group and Europe organization for research and treatment of cancer late radiation morbidity scoring scheme
Loco regional control rates (LCR) | 3-5 years
  Defined as the time from the date of randomization to 1st failure in nasopharynx or neck lymph nodes
Progression free survival (PFS) | 3-5 Years
  Defined as the time from the date of randomization to 1st failure locally or systemically

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Defined as the time from the date of randomization to death from any cause
Distance Metastasis free survival (DMFS) | 5 years
  It is evaluated and calculated from the date of random assignment until date of first distance metastasis or until the date of last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Issa, MD, Principal Investigator — KCCC
Locations (1):
- Kuwait Cancer Control Center, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Lee AW, Sze WM, Au JS, Leung SF, Leung TW, Chua DT, Zee BC, Law SC, Teo PM, Tung SY, Kwong DL, Lau WH. Treatment results for nasopharyngeal carcinoma in the modern era: the Hong Kong experience. Int J Radiat Oncol Biol Phys. 2005 Mar 15;61(4):1107-16. doi: 10.1016/j.ijrobp.2004.07.702. PMID 15752890
- [Background] Al-Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol. 1998 Apr;16(4):1310-7. doi: 10.1200/JCO.1998.16.4.1310. PMID 9552031
- [Background] Langendijk JA, Leemans CR, Buter J, Berkhof J, Slotman BJ. The additional value of chemotherapy to radiotherapy in locally advanced nasopharyngeal carcinoma: a meta-analysis of the published literature. J Clin Oncol. 2004 Nov 15;22(22):4604-12. doi: 10.1200/JCO.2004.10.074. PMID 15542811
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014
- See also: Globocan.fr. Accessed January 2020. — https://gco.iarc.fr/
- See also: chemotherapy protocols — http://www.bccancer.bc.ca/health-professionals/clinical-resources/cancer-drug-manual/drug-index